CLINICAL TRIAL: NCT06635382
Title: Clinical Evaluation of Dimethyl Sulfoxide Wet Bonding Technique: A Randomized Controlled Trial
Brief Title: Clinical Evaluation of Dimethyl Sulfoxide Wet Bonding Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manipal University College Malaysia (Other)
Responsible Party: Principal Investigator, Philip Pradeep, Associate Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 049/2023
Record Dates: First submitted 2024-09-02; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Dimethyl Sulfoxide
MeSH Terms: interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Universal single bond adhesive (Active Comparator)
  Interventions: Other: Universal single bond adhesive
- DMSO application before Universal single bond adhesive (Experimental)
  Interventions: Other: Universal single bond adhesive; Other: DMSO

INTERVENTIONS:
Other: Universal single bond adhesive — Will be applied and light cured for 20 seconds.
Other: DMSO — DMSO application on tooth followed by active application of universal single bond adhesive and light cured for 20 seconds.
  Arms: DMSO application before Universal single bond adhesive

SUMMARY:
Dimethyl sulfoxide (DMSO) wet bonding has shown promising results in several in vitro studies. However, there are a lack of clinical trials which prove the advantages of this technique. The aim of the study is to clinically assess the effect of DMSO wet bonding on composite restoration in non carious cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

* Two similar non carious cervical lesions (NCCLs) on the facial/labial surfaces of premolars.
* NCCLs of score 1-3 on the Smith and Knight tooth wear index.
* Favorable occlusion and teeth are in normal contact.

Exclusion Criteria:

* NCCLs on the lingual surface.
* Medically compromised individuals.
* Periodontally compromised teeth.
* Bruxism and visible wear facets in the posterior dentition.
* Fractured or visibly cracked premolars and canines.
* Known allergies to resin-based restorative materials.
* Presently undergoing orthodontic treatment.
* Abutment teeth for fixed or removable prostheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Fracture of material | From treatment to 3-6 months follow up
  Different fracture patterns and retention failures may occur in relation to the type of restoration: cracks, chipping/ delamination, bulk fractures, or incomplete and complete loss of retention. Assessed by Visual examination and short air drying. Criteria set from Clinically excellent/very good(sufficient) (Score 1) to Clinically poor (entirely insufficient)(Score 5)
Marginal adaptation | From treatment to 3-6 months follow up
  There are different interfaces between the dental hard tissue, restorative material, and adhesive and/or luting resin/cement layer. Each interface can degrade and potentially alter marginal adaptation. In clinical practice, it is impossible to distinguish failures between the different interfaces. Therefore, only the marginal adaptation as such can be assessed by visual examination and short air drying.
  Scores given depending upon the quality of restoration from Clinically excellent/very good (sufficient) (Score 1) to Clinically poor (entirely insufficient) (Score 5)

REFERENCES:
- [Result] Lopez-Frias FJ, Castellanos-Cosano L, Martin-Gonzalez J, Llamas-Carreras JM, Segura-Egea JJ. Clinical measurement of tooth wear: Tooth wear indices. J Clin Exp Dent. 2012 Feb 1;4(1):e48-53. doi: 10.4317/jced.50592. eCollection 2012 Feb. PMID 24558525
- [Result] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246